CLINICAL TRIAL: NCT04151368
Title: Robotic Nipple-Sparing Mastectomy With Immediate Prosthetic Breast Reconstruction: Prospective Study of Feasibility, Safety and Patient Satisfaction, Toronto Experience.
Brief Title: Surgical and Patient Reported Outcomes of Robotic Nipple-Sparing Mastectomy
Acronym: RNSM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been temporarily suspended since the start of the pandemic due to the need for travel for this study. Will resume when appropriate.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-5250.0
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Surgery--Complications; Genetic Predisposition to Disease; Surgery; BRCA1 Mutation; BRCA2 Mutation; Breast Diseases
Keywords: breast surgery; robotic surgery; nipple sparing mastectomy; genetic predisposition; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease; Breast Diseases

STUDY DESIGN:
Intervention Model Description: Prospective Single Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Robotic Nipple Sparing Mastectomy Arm (Experimental): Patient cohort undergoing nipple sparing mastectomy with use of robotic dissection.
  Interventions: Procedure: Robotic Nipple-Sparing Mastectomy (RNSM)

INTERVENTIONS:
Procedure: Robotic Nipple-Sparing Mastectomy (RNSM) — RNSM will be performed by previously described method using 3 cm extra-mammary axillary incision along the mid-axillary line in the axillary fossa. We will use Da Vinci Si Surgical System® (Intuitive Surgical, Sunnyvale, CA).

SUMMARY:
Nipple-sparing mastectomy (NSM) with immediate reconstruction is one of the standard of care surgical treatments of breast cancer (BC) and is used for risk reduction in patients with a high risk for BC. While this method shows satisfactory oncologic and good cosmetic outcomes, its drawbacks include compromise of the skin flap vascularization due to skin incision, nipple-areolar complex (NAC) malposition/distortion and visible scar on the breast. NSM also has technical challenges of dissecting and removing larger specimens through limited incisions and concerns regarding oncologic effectiveness due to difficulties in visualizing regions of the breast remote from the incision. To improve cosmetic outcomes after NSM, a modification of this technique using a surgical robotic system was recently described. In a limited number of studies, the robotic NSM (RNSM) with immediate prosthetic breast reconstruction (IPBR) was shown to be feasible and safe, as well as led to excellent cosmetic outcomes and patient satisfaction. There are limited number of centers in North America and none in Canada that offer RNSM-IPBR. The investigators hypothesize that RNSM-IPBR is a feasible and safe technique that can be utilized in our institution and that it can provide superior cosmetic outcomes with less morbidity and higher patient satisfaction compared to the traditional NSM-IPBR. The aim is to conduct a single-arm prospective study to investigate the safety and feasibility, as well as cosmetic, surgical complication and patient satisfaction parameters of NSM-IPBR performed in the University Health Network (UHN). This study will serve a foundation for potential introduction of a novel surgical approach in our institution and will make it available for treatment and prevention of breast cancer in Canadian women. The study will also serve as pilot data for future potential studies, including randomized-controlled trials (RCT) comparing RNSM with conventional NSM. As such, the study will further our approach to innovation in breast surgical oncology within Canada and North America.

DETAILED DESCRIPTION:
This is a single-arm prospective study to assess feasibility and safety (primary outcomes), as well as patient satisfaction, cosmetic and oncologic outcomes of RNSM-IPBR in women with BC or at high risk of BC treated at UHN.

The objectives of the study are to determine:

1. Feasibility of RNSM-IPBR through assessing operative parameters (such as time of procedure, robot docking time, conversion to conventional NSM-IPBR).
2. Safety of RNSM-IPBR through assessing rate of morbidity from surgical complications (such as wound infection, flap and NAC necrosis, postoperative hematoma/bleeding, seroma requiring aspiration, implant loss, anesthesia related complications and need for reoperation with one month due to complications) and mortality due to the procedure.
3. Patient satisfaction from RNSM-IPBR through assessing psychological, physical, sexual well-being, as well as satisfaction with breast, overall outcome and care through patient reported outcomes.
4. Cosmetic outcomes of RNSM-IPBR, such as distortion or malposition of NAC and scarring, rate of reoperation due to unacceptable cosmetic outcomes.
5. Short- and long-term oncologic outcomes of NSM-IPBR, such as positivity of margins, breast cancer incidence and recurrence rate, as well as overall survival.

The rationale of the study is to investigate a novel technique of RNSM-IPBR that might have superior cosmetic and patient satisfaction outcomes, as well as lower rates of complications, based on a small number of previously published studies from Europe and Asia.

Once enrolled, clinical, radiologic, and pathologic data will be collected for each participant at the initial visit and follow up data will be collected via available electronic patient records.

RNSM-IPBR will be performed by previously described method (Toesca et al.) using an extra-mammary axillary incision along the mid-axillary line in the axillary fossa. We will use Da Vinci Si Surgical System® (Intuitive Surgical, Sunnyvale, CA) available at Toronto General Hospital, UHN.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age with invasive breast cancer (BC), ductal carcinoma in situ (DCIS), BRCA or other breast cancer genetic mutation carriers or high risk BC female patients who are otherwise candidates for NSM with IPBR will be eligible for the study. For those patients, RNSM-IPBR will be offered. Those who, after thorough discussion of risks and benefits, choose and consent to undergo RNSM-IPBR will be included in the study.

Exclusion Criteria:

* Heavy smokers (>20 cigarettes a day)
* Uncompensated Diabetes Mellitus
* High risk for anesthesia (ASA 4)
* Inflammatory Breast Cancer
* Previous thoracic radiation therapy for any reason
* Pregnancy
* Psychiatric, addictive, or any disorder which compromises ability to give informed consent for participation in this study

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with increased lifetime risk of breast cancer Female patients with early stage breast cancer
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of RNSM | 1 month
  Surgical time in minutes
Wound complications | 2 months
  Skin and Nipple necrosis
Margins after RNSM | 1 month
  Margin status (mm)
Breast cancer recurrence | 36 months
  Site of first relapse

SECONDARY OUTCOMES:
Patient Satisfaction | Pre-Operative and 6 and 12 months post-operative
  Breast Q Pre and Post-operative Surveys- items measuring satisfaction with appearance, surgical experience, breast shape and symmetry, psychosocial, physical and sexual well being. Lowest score = 0, highest = 100 with higher scores indicating better outcomes / quality of life.
Body Image | 6 months post-operative
  Hopwood's Body Image Scale- Scores range from 0 (min distress) to 3 (max distress) for 10 questions. Lowest score = 0, highest = 30 with lower scores indicated lower body image distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tulin D Cil, MD, MEd, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Background] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Tran de Fremicourt K, Conversano A, Rimareix F, Simon M, Michiels S, Kolb F. Robotic Prophylactic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: A Prospective Study. Ann Surg Oncol. 2018 Sep;25(9):2579-2586. doi: 10.1245/s10434-018-6555-x. Epub 2018 Jun 29. PMID 29959612